CLINICAL TRIAL: NCT07078240
Title: "You Sure or Not?" Examining the Trust, Acceptance and Adoption of Falls Risk - Artificial Intelligence Recommender (FAIR) System by Nurses
Brief Title: Examining Nurses' Trust and Acceptance of FAIR, an AI-powered Falls Risk Recommender
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Marquette University (Other); Lee Kong Chian School of Medicine, Nanyang Technological University (Unknown)
Responsible Party: Principal Investigator, Glass George Frederick Jr, Deputy Head of Nursing Research, Tan Tock Seng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRCRTF25jan-004
Record Dates: First submitted 2025-06-22; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Falls Risk
Keywords: Artificial Intelligence trust; Artificial Intelligence acceptance; Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: Two phases of interventional study. First is a parallel arm study comparing nurse acceptance and trust in intervention vs control arm in simulation lab setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Nurses in the intervention arm will perform will receive training on the nature of AI recommender (FAIR) and how it works, and how they can apply it in their assessment of the patient.
  After that, they will be introduced to three simulated patients with different conditions and needs - intended to reflect a patient at "low risk of falls", "moderate risk of falls" and "high risk of falls" and asked to read and interpret the FAIR recommendations before making their own falls risk assessment of the patient using mWHeFRA.
  Interventions: Other: Falls risk - Artificial Intelligence Recommender (FAIR)
- Control arm (Placebo Comparator): Nurses in the control arms will be reinforced on fall risk assessment methods using the modified Western modified Western Health Falls Risk Assessment Tool (mWHeFRA).
  After that, they will be introduced to three simulated patients with different conditions and needs - intended to reflect a patient at "low risk of falls", "moderate risk of falls" and "high risk of falls" and asked to perform assessments of the patient mWHeFRA.
  Interventions: Other: modified Western Health Falls Risk Assessment Tool (mWHeFRA)

INTERVENTIONS:
Other: Falls risk - Artificial Intelligence Recommender (FAIR) — FAIR is an alert system built into the hospital's electronic medical record system. It is an adaptation of a machine learning model for fall risk calculation built in another hospital in Singapore. FAIR combines multiple patient-specific variables to identify if a patient is at increased risk of falling during their inpatient stay, marking them as a 'falls risk'.
  Based on the 'flag' raised, the nurse will be instructed to prioritise her falls risk assessment of the patient (If deemed 'high risk') or to do so subsequently as a lower priority once other pressing patient care issues are resolved (if deemed 'low risk').
  That way, it ensures the requirements of each patient receiving a falls risk assessment as scored through mWHeFRA are still met, with FAIR allowing nurses to better prioritise their focus and attention on the patient that most needs the assessment at point of admission,
  Arms: Intervention Arm
Other: modified Western Health Falls Risk Assessment Tool (mWHeFRA) — The mWHeFRA is the hospital's standard falls risk assessment tool. All nurses are expected to be proficient in its use to guide their risk assessment of patients
  Arms: Control arm

SUMMARY:
An exploratory mixed-method study will be conducted to test acceptance and trust of an AI-powered falls risk predictor system by inpatient hospital nurses

DETAILED DESCRIPTION:
This protocol covers the trial component of a 4-year PhD research study covering focus group discussions with nurses on AI risk systems, workshops to gather feedback on the AI system and feasibility testing in a simulated environment and clinical environment

ELIGIBILITY:
Inclusion Criteria:

* Practicing nurse involved in falls risk assessments of patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of FAIR's flag acceptance | 1 Day of Study
  Examination of how often the flags raised by FAIR are accepted by nurses, and whether they are accepted or ignored correctly.
Time taken to do falls risk assessment | 1 Day of Study
  The time taken by the nurses to perform their falls risk assessment will be recorded

SECONDARY OUTCOMES:
Time spent looking at FAIR | 1 Day of Study
  The time each nurses takes looking at the FAIR falls risk assessment will be assessed
Baseline and Post-Simulation Nurse trust and acceptance of FAIR | Baseline
  Measured by the adapted Unified Theory of Acceptance and Use of Technologies and System Usability Survey, adjusted to better capture the key predictors of nurse acceptance

IPD SHARING:
Plan to Share IPD: Yes
Will be agreeable to share Protocol Summary page
Time Frame: Available from 2026 to 2036
Access Criteria: Individuals will have to contact me as Primary Investigator for permission to use

REFERENCES:
- [Background] Schulz PJ, Lwin MO, Kee KM, Goh WWB, Lam TYT, Sung JJY. Modeling the influence of attitudes, trust, and beliefs on endoscopists' acceptance of artificial intelligence applications in medical practice. Front Public Health. 2023 Nov 28;11:1301563. doi: 10.3389/fpubh.2023.1301563. eCollection 2023. PMID 38089040